CLINICAL TRIAL: NCT02463110
Title: Acute Myocardial Necrosis and Depression: Antiplatelet Effect of Reuptake Inhibition of Serotonin: The ANDROS Study
Brief Title: Acute Myocardial Necrosis and Depression: Antiplatelet Effect of Reuptake Inhibition of Serotonin
Acronym: ANDROS
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Investigator's decision
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Action Research Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P110155
Record Dates: First submitted 2015-05-19; First posted 2015-06-04 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-05

CONDITIONS: Depression; Coronary Artery Disease
Keywords: Acute Coronary Syndrome; Depression; Coronary Artery Disease; Myocardial Infarction; Percutaneous Coronary Intervention
MeSH Terms: conditions — Depression; Coronary Artery Disease; Acute Coronary Syndrome; Myocardial Infarction | interventions — Sertraline; WW Domain-Containing Oxidoreductase

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1: Sertraline (Experimental): ACS, depression
  Interventions: Drug: Sertraline
- 2: Placebo (Placebo Comparator): ACS, depression
  Interventions: Drug: Placebo
- 3: Control (Other): ACS, no depression, no treatment
  Interventions: Drug: No treatment

INTERVENTIONS:
Drug: Sertraline — Sertraline one capsule (50mg per day), which can be increased up to 200mg per day (maximum dose) for 6 months.
  Arms: 1: Sertraline
Drug: No treatment
  Arms: 3: Control
Drug: Placebo
  Other Names: Placebo one capsule, which can be increased up to 4 capsules per day (maximum dose) for 6 months.
  Arms: 2: Placebo

SUMMARY:
Primary purpose:

To evaluate the evolution in time of the antiaggregant platelet effect of sertraline (SSRI) compared to placebo in depressive patients with ACS (Acute Coronary Syndrome) and treated as recommended by a double antiplatelet therapy, aspirin and clopidogrel.

Hypothesis:

The benefits of SSRIs observed in depressive patients with ACS are related to an antiplatelet effect.

DETAILED DESCRIPTION:
Rational:

40% of patients hospitalized for acute coronary syndrome (ACS) present depressive symptoms. The increase in cardiovascular morbidity and mortality at 6 months (hazard ratio = 3.5) could partly be explained by an alteration of the platelet parameters in patients with depression.

Sertraline is a potent inhibitor of the selective serotonin reuptake (SSRI). At the platelet level, it decreases the secretion induced by collagen and causes the inhibition of serotonin reuptake and platelet activation, wider than the simple anti-serotonergic effect. Its efficacy on depression of patients with ACS has been demonstrated (-20% of ischemic events at 24 weeks vs placebo), partly independent of the correction of depressive symptoms, and with a wide safety action. Antiplatelet, anti-inflammatory and endothelial function effects of sertraline are demonstrated in healthy volunteers, in stable patients and in patients with heart failure, but have never been explored in ACS .

Multicenter, randomized, double-blind, controlled trial comparing SSRI and placebo in depressive patients with ACS.

A control (non depressive) ACS group will also do the clinical and laboratory follow-up at the same time (without drug administration), to constitute a reference for platelet parameters and to allow a comparison with the depressive ACS group treated with placebo.

Randomization and initiation of the treatment at the end of the hospitalization for ACS (possibly after reperfusion and stabilization of cardiac medication)

ELIGIBILITY:
Inclusion Criteria:

* Patient Aged 18 years and older
* Patient Depressive without antidepressant therapy for three months (valid only for the sertraline and placebo groups)
* Patient With ACS with elevated cardiac enzymes (above the 99th percentile of the upper limit of normal of the laboratory)
* Patient That assessed depressive symptoms : Test Beck (13 items)
* Patient Affiliated to a social security scheme (beneficiary or assignee)
* Patient Having signed a free and informed consent

Exclusion Criteria:

* Cardiovascular

  * History of serious bleeding (recent hemoglobin fall 5g / dl ( <3 months ), intracranial hemorrhage or hemorrhagic tamponade)
  * Uncontrolled hypertension (SBP > 180 mmHg or DBP > 100 mmHg)
  * Stroke <3 months
  * Treatment with ticagrelor or prasugrel for the duration of the study.
* Psychiatric

  * Psychosis, bipolar illness
  * Dementia (Mini- Mental State Examination score < 23)
  * Uncontrolled epilepsy
  * Severe depression (score > 15) with suicidal risk identified by a psychiatrist (urgent treatment for depression needed)
  * Patient experienced depression and treated in the last three months or currently receiving treatment
  * Treatment with selective and non-selective monoamine oxidase inhibitors of the group A within 14 days prior to the introduction of sertraline
* Clinical and Biological

  * Prothrombin time > 1.5 second
  * Platelet rate < 100 000 / mm3
  * Hematocrit rate < 25%
  * Serum creatinine > 4.0 mg / dl
  * Severe hepatic impairment (Child Pugh stage C)
* Contraindications to sertraline (placebo / sertraline group)

  * Hypersensitivity to the active substance or to any of the excipients (anhydrous lactose, pregelatinized corn starch, sodium laurilsulfate , magnesium stearate)
  * Treatment with pimozide
  * Genetic galactose intolerance, malabsorption of glucose and galactose, lactase deficiency
* Regulatory

  * Women without effective contraception or pregnant or lactating or desiring pregnancy or within 6 months after randomization
  * Participation in biomedical research on other drugs during the period of participation
  * Patients unable to follow the treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-07; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Time dependent pattern of changes in platelet reactivity under sertraline compared to placebo within a time Frame of 6 months of treatment | 0 day, 1 day, 6 weeks, 24 weeks, 28 weeks
  To evaluate the time variation of the level of platelet reactivity (ADP induced residual aggregation) under sertraline compared to placebo within a time Frame of 6 months of treatment.
  Time Frame:
  T0 = before starting treatment with sertraline T1 = at discharge from the hospital = J1 after introduction of treatment with sertraline T2 = 6 weeks of treatment with sertraline T3 = 24 weeks of treatment with sertraline = end of treatment with sertraline T4 = 4 weeks after the end of treatment with sertraline (biological and psychiatric rebound)

SECONDARY OUTCOMES:
Time dependent pattern of changes in platelet activation | 0 day, 1 day, 6 weeks, 24 weeks, 28 weeks
  Maximal platelet aggregation (ADP, Arachidonic Acid, Collagen), markers of platelet activation (betaTG, CD40s)
Time dependent pattern of changes in inflammation markers | 0 day, 1 day, 6 weeks, 24 weeks, 28 weeks
  Dosage of inflammation markers (IL-6, CRP, Fg, myeloperoxydase)
Time dependent changes in Depression | 0 day, 1 day, 6 weeks, 24 weeks, 28 weeks
  Beck Depression Inventory (BDI)
Time dependent changes in Tobacco addiction | 0 day, 1 day, 6 weeks, 24 weeks, 28 weeks
  Fargenström test
Time dependent changes in Bleeding risk | 0 day, 1 day, 6 weeks, 24 weeks, 28 weeks
  Dosage of hemoglobin, hematocrit and follow-up of hemorrhage

CONTACTS AND LOCATIONS:
Overall Officials: Johanne SILVAIN, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- ACTION Group - Pitié-Salpêtrière University Hospital (APHP), Paris, France